CLINICAL TRIAL: NCT01059240
Title: SMN Copy Number Distribution in Mali, West Africa
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999910033; 10-N-N033
Record Dates: First submitted 2010-01-28; First posted 2010-01-29 (Estimated); Last update posted 2019-12-05 (Actual); Status verified 2017-05-18

CONDITIONS: Spinal Muscular Atrophy
Keywords: Survival Motor Neuron 1 (SMN1); Survival Motor Neuron 2 (SMN2); Spinal Muscular Atrophy (SMA); SMN Copy Number in Mali; Spinal Muscular Antrophy; SMA
MeSH Terms: conditions — Muscular Atrophy, Spinal

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Background:

* Spinal muscular atrophy (SMA) is a degenerative and incurable neuromuscular disorder that is caused by mutations in the survival motor neuron gene, SMN1, found on chromosome 5. It is the leading inherited cause of infant mortality. SMA carriers (those who have the genetic mutation but do not have the disease) are often unaware of their status until they are tested.
* Researchers have been studying the prevalence of SMA carriers in the general population, but most of the information collected has come from populations within the United States, Europe, and Asia. Very few studies have been performed in Africa. Furthermore, this information does not provide much information regarding carrier frequency based on ethnic background and ancestry. To address this problem, researchers are interested in studying the prevalence of the SMA genetic mutation in the sub-Saharan nation of Mali.

Objectives:

- To collect blood samples for use in studying genetic data related to spinal muscular atrophy.

Eligibility:

* Healthy volunteers who are at least 18 years of age.
* Volunteers will be of Malian ancestry and nationality.

Study Location:

-<TAB>Bamako, Mali, West Africa

Design:

* The study will first collect blood samples from a small group of volunteers to run initial SMA carrier testing and resolve any technical difficulties before continuing with the study.
* Participants will complete questionnaires about their personal and family medical history, including questions about illnesses, stillborns, and miscarriages, and then will provide blood samples for genetic research and testing.

DETAILED DESCRIPTION:
Objective

Spinal muscular atrophy (SMA) is an autosomal recessive motor neuron disease that is caused by mutations in the survival motor neuron gene, SMN1. The objective of this study is to determine the SMN copy number distribution in the Malian population and to compare this to published data obtained elsewhere. It is anticipated that this study will help to refine the knowledge of SMA by assessing the distribution of SMN copy number, and the SMA carrier frequency in a sub-Saharan nation, thus expanding the information base available to clinicians and patients considering SMA carrier testing.

Study Population

The study population will include 1400 adult (18 years of age and older) volunteers only.

Design

Blood samples from volunteers will be collected from students at the School of Medicine, Pharmacy, and Dentistry (FMPOS) at the University of Bamako, which consists of an ethnically diverse population representative of the Malian ethnicities. No therapy will be provided to study participants.

Outcome Measures

Outcome measure for phase 1 is DNA extraction yield of sufficient quantity and quality for SMN genotyping by LabCorp in at least 90% of samples. Outcome measures for phase 2 are the frequency of SMA carriers (SMN1 deletion heterozygotes) and the SMN1 and SMN2 copy number distribution in Mali.

Abbreviations and Definition of Terms

* SMA: Spinal Muscular Atrophy
* SMN: Survival Motor Neuron
* SMN1: Survival Motor Neuron Telomeric
* SMN2: Survival Motor Neuron Centromeric

ELIGIBILITY:
* INCLUSION CRITERIA:

Medical students at the FMPOS of Malian ancestry and nationality who are 18 years of age and above will be considered for this study.

EXCLUSION CRITERIA:

Subjects may not be eligible to participate if they have a condition that would make a single 6 ml blood draw unsafe. Student assistants are ineligible for the study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 701 (Actual)
Dates: Start 2010-01-21; Study Completion 2017-05-18

PRIMARY OUTCOMES:
Primary outcome measure for phase 1 is DNA extraction yield of sufficient quantity and quality for SMN genotyping in at least 90% of samples

SECONDARY OUTCOMES:
Secondary outcome measures for phase 2 are the frequency of SMA carriers (SMN1 deletion heterozygotes) and the SMN1 and SMN2 copy number distribution in Mali.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth H Fischbeck, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- University of Bamako, Faculty of Medicine, Pharmacy and Dentistry (FMPOS), Bamako, Mali

REFERENCES:
- [Background] Lefebvre S, Burlet P, Liu Q, Bertrandy S, Clermont O, Munnich A, Dreyfuss G, Melki J. Correlation between severity and SMN protein level in spinal muscular atrophy. Nat Genet. 1997 Jul;16(3):265-9. doi: 10.1038/ng0797-265. PMID 9207792
- [Background] Smith M, Calabro V, Chong B, Gardiner N, Cowie S, du Sart D. Population screening and cascade testing for carriers of SMA. Eur J Hum Genet. 2007 Jul;15(7):759-66. doi: 10.1038/sj.ejhg.5201821. Epub 2007 Mar 28. PMID 17392705
- [Background] Wirth B, Schmidt T, Hahnen E, Rudnik-Schoneborn S, Krawczak M, Muller-Myhsok B, Schonling J, Zerres K. De novo rearrangements found in 2% of index patients with spinal muscular atrophy: mutational mechanisms, parental origin, mutation rate, and implications for genetic counseling. Am J Hum Genet. 1997 Nov;61(5):1102-11. doi: 10.1086/301608. PMID 9345102